CLINICAL TRIAL: NCT00404144
Title: PEPCAD I, The Paclitaxel-Eluting PTCA-Balloon Catheter to Treat Small Vessel Coronary Artery Disease. A Pilot Study
Brief Title: PEPCAD I. The Paclitaxel-Eluting PTCA-Balloon Catheter to Treat Small Vessel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heart Centre Rotenburg (Other)
Collaborators: B. Braun Melsungen AG (Industry); Clinical Research Institute, Center for Cardiovascular Disease Rotenburg a.d.F. (Unknown)
Responsible Party: Principal Investigator, Ralf Degenhardt, PhD, Data Manager, Heart Centre Rotenburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID: BBM-VS-52; PEPCAD II/CRI/05/-01/c-c
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Stenosis
Keywords: small vessel; paclitaxel coated balloon catheter; pepcad; drug eluting balloon
MeSH Terms: conditions — Coronary Stenosis

ARMS (1):
- Drug Eluting Balloon (Experimental): treatment of small vessel with drug eluting balloon
  Interventions: Device: Drug Eluting Balloon

INTERVENTIONS:
Device: Drug Eluting Balloon — PCI of small vessels single arm study

SUMMARY:
The objective of this study is to assess the safety and efficacy of the Paclitaxel-eluting PTCA-balloon catheter (3µg/mm2 balloon surface area) in the treatment of significant (≥ 70% and < 100 %) stenoses in native coronary arteries with reference diameters from 2.25 mm to 2.8 mm and ≤ 22 mm in length for procedural success and preservation of vessel patency.

DETAILED DESCRIPTION:
Background information:

Stent deployment for the treatment of coronary artery stenoses has evolved as the standard treatment in nearly all types of coronary lesions over the past two decades. The initial recurrence rate of bare stents in the range of 20 30 % in low risk stenoses has been further reduced by devices with passive coatings such as silicon carbide, heparin, phosphorylcholine, and carbon.

In the percutaneous transluminal treatment of stenotic coronary arteries with diameters below 3 mm, however, none of the currently available methods, namely balloon angioplasty with conventional balloons (POBA) and deployment of non-drug eluting stents have shown acceptable results for the various reasons inherent to these approaches. Although some studies showed POBA and the deployment of bare stents to be equally effective with respect to restenosis, in a recently published meta-analysis of eleven trials the restenosis rates were as high as 25.8 % for POBA and 34.2 % for bare stents, respectively.

Brachytherapy initially demonstrated encouraging results. However, due to its disadvantages such as delayed endothelialization, the risk associated with additional stenting, the cumbersome logistics at the sites and in the labs, brachytherapy is not considered as a valid approach. Data with the Sirolimus-eluting Cypher™ stent in vessels averaging 2.60 ± 0.54 mm in diameter showed the benefit of this cytostatic drug in this indication. However, this approach introduces a layer of metal to the per se small vessel and, thus, reduces the vascular lumen.

Study Rationale:

Since none of the above mentioned options for the percutaneous treatment of small vessel coronary artery stenoses seems to be universally recommendable the Paclitaxel-eluting PTCA balloon catheter has to be considered as an alternative. The possible advantages over either the uncoated balloon or bare stent include the antiproliferative mode of action of the compound. In comparison to the drug eluting stents (DES) the homogenous distribution of the compound along the target vessel segment, the lack of chronic mechanical alteration of the artery and the ease of access to the lesion would favor the Paclitaxel-eluting balloon.

However, there are no data available on the use of the drug eluting balloons in small vessel disease and the information on the other indication evaluated to date, the treatment of in-stent restenosis is limited. In the latter indication, the animal model and according to unpublished results in humans, the proliferation induced by a Paclitaxel-eluting balloon catheter was significantly less compared to an uncoated balloon, the Paclitaxel-coated Taxus™ stent, and to the Sirolimus-eluting Cypher™ stent. Therefore, it is prudent to test the Paclitaxel-eluting PTCA balloon catheter as an alternative approach for the percutaneous transluminal treatment of small vessel coronary artery lesions.

Since none of the alternative methods has unequivocally shown its superiority over the other, none of them may serve as the golden standard and, i.e., for direct comparison. Consequently, as the initial step conducting a single arm study with the Paclitaxel-eluting balloon is suggested with historic data serving for comparison. Once these results will have been obtained a prospective randomized trial shall be discussed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable angina pectoris (CCS class 1-3) or with unstable angina pectoris (Braunwald class 1-2, A-C) or documented ischemia or with documented silent ischemia
* Patients eligible for coronary revascularization by means of PCI
* Patients suitable for coronary revascularization of any sort (balloon angioplasty, device-assisted balloon-angioplasty or coronary artery bypass grafting)
* Women of childbearing potential may not be pregnant nor have the desire to becoming pregnant during the first year following the study procedure. Hence, patients will be advised to use an adequate birth control method up to and including 6 months follow-up.
* Patients who are mentally and linguistically able to understand the aim of the study and to show sufficient compliance in following the study protocol
* Patients must agree to undergo the 6 months angiographic follow-up
* Patients must agree to undergo the 1 and 3 year clinical follow-up
* Patient is able to verbally acknowledge an understanding of the associated risks, benefits, and treatment alternatives to therapeutic options of this trial, e.g., balloon angioplasty by means of the Paclitaxel-eluting PTCA-balloon catheter. The patients, by providing their informed consent, agree to these risks and benefits as stated in the patient informed consent document
* Patients with medical indication for follow-up angiography
* Reference diameters from 2.25 mm to 2.8 mm and ≤ 22 mm in length
* Diameter stenosis pre procedure must be either > 70 % or >50 % if ischemia corresponding to the target lesion is documented either by exercise stress ECG, stress echocardiography, or scintigraphy
* The target lesion must be covered by a single Paclitaxel-eluting balloon

Exclusion Criteria:

* Patients with acute (< 24 h) or recent (≤ 48 hours) myocardial infarction
* Patients with unstable angina pectoris (Braunwald class 3)
* Patients with severe congestive heart failure
* Patients with severe heart failure NYHA IV
* Patients demonstrating clinical signs of cardiogenic shock at the time of the procedure (systolic blood pressure of less than 80 mm Hg requiring inotropic support, IABP and/or fluid challenge).
* Women who are pregnant or lactating
* Patients with another coronary stent implanted previously into the target vessel
* Patients with bleeding diathesis in whom anticoagulation or anti-platelet medication is contraindicated
* Patient participates in other clinical trials involving any investigational device or drug
* Untreated hyperthyroidism
* Patient has presence or history of severe renal failure (GFR<30ml/min) and is therefore not eligible for angiography. Patient's serum creatinine levels must be documented
* Post transplantation of any organ or immune suppressive medication
* Other disease to jeopardize follow-up (e.g., malignoma)
* Addiction to any drug or to alcohol
* Patients with any type of surgery during the week preceding the interventional procedure
* Evidence of extensive thrombosis within target vessel before the intervention
* Side branch > 2 mm in diameter originating from the lesion
* Bifurcate lesion
* Restenotic lesion
* Multilesion percutaneous coronary intervention within the same artery (a main artery (e.g., LCdx) and its side branch (e.g., OMS) are considered as different arteries)
* Percutaneous coronary intervention of venous graft
* Target segment is occluded (i.e., acute or chronic)
* In-stent restenosis
* Ostial lesion within 2 mm of vessel origin
* Patient is intolerant to aspirin and/or the ADP-antagonists clopidogrel or has a history of neutropenia, thrombocytopenia induced by ADP-antagonists, or severe hepatic dysfunction prohibiting the use of clopidogrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-01; Primary Completion 2010-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Late lumen loss at 6 months | 6 month

SECONDARY OUTCOMES:
Procedural success | during procedure
30-day MACE rate | 30 days
Percent stenosis at 6 months | 6 months
Binary restenosis rate at 6 months | 6 months
Late loss index at 6 months | 6 months
Cumulative MACE rate at 6 months | 6 months
Cumulative MACE rate at 1 year | 1 year
Cumulative MACE rate at 3 years | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: M. Unverdorben, MD,PhD, Principal Investigator — Center for Cardiovascular Diseases, Heinz-Meise-Strasse 100, D-36199 Rotenburg a.d. Fulda, Germany
Locations (9):
- Germany (9):
  - Kerckhoff-Clinic Bad Nauheim, Bad Nauheim
  - Unfallkrankenhaus Berlin, Berlin
  - Medizinische Klinik, Kardiologie, St.-Johannes -Hospital, Dortmund
  - Städtische Kliniken Esslingen, Klinik für Kardiologie, Angiologie und Pneumologie, Esslingen am Neckar
  - Martin-Luther-Universität Halle-Wittenberg, Universitätsklinik und Poliklinik für Innere Medizin III, Halle
  - University of Heidelberg, Clinic for Internal Medicine, Dept. of Cardiology, Heidelberg
  - University of Saarland, Internal Medicine III, Homburg/Saar
  - Universitätklinikum Jena, Klinik für Innere Medizin, Jena
  - Center for Cardiovascular Diseases, Cardiologic Clinic, Rotenburg A.d. Fulda

REFERENCES:
- [Derived] Unverdorben M, Kleber FX, Heuer H, Figulla HR, Vallbracht C, Leschke M, Cremers B, Hardt S, Buerke M, Ackermann H, Boxberger M, Degenhardt R, Scheller B. Treatment of small coronary arteries with a paclitaxel-coated balloon catheter in the PEPCAD I study: are lesions clinically stable from 12 to 36 months? EuroIntervention. 2013 Sep;9(5):620-8. doi: 10.4244/EIJV9I5A99. PMID 24058078
- [Derived] Unverdorben M, Kleber FX, Heuer H, Figulla HR, Vallbracht C, Leschke M, Cremers B, Hardt S, Buerke M, Ackermann H, Boxberger M, Degenhardt R, Scheller B. Treatment of small coronary arteries with a paclitaxel-coated balloon catheter. Clin Res Cardiol. 2010 Mar;99(3):165-74. doi: 10.1007/s00392-009-0101-6. Epub 2010 Jan 6. PMID 20052480